CLINICAL TRIAL: NCT01792895
Title: Is Better the One Type of Manual Therapy Than Others for to Treat the Patients With Chronic Neck Pain? : A Randomized Clinical Trial
Brief Title: Different Types of Manual Therapy Techniques in Patients With Chronic Neck Pain
Acronym: CNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD and Physical Therapist, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A04-12
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Neck Pain
Keywords: Posterior Neck Pain; Cervical spine pain; Manual therapy
MeSH Terms: conditions — Neck Pain | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Manipulation group (Active Comparator): This Technique will be applied over four sessions, during two weeks
  Interventions: Procedure: Mobilization; Procedure: Mobilization with movement
- Mobilisation (Active Comparator): This treatment will be applied on cervical spine during four sessions, over two weeks
  Interventions: Procedure: Manipulation; Procedure: Mobilization with movement
- Mobilization with movement (Active Comparator): This Technique will be applied over four sessions, during two weeks
  Interventions: Procedure: Manipulation; Procedure: Mobilization

INTERVENTIONS:
Procedure: Manipulation — The Cervical Spine Manipulation is a manual therapy technique directed at the hypomobile and painful vertebral level. The subject was supine with the cervical spine in a neutral position. The index finger of the therapist applies contact over the posterolateral aspect of the zygapophyseal joint of the hypomobile vertebra. The therapist performs the technique taking account the most limited movement; lateral or rotational. A maximum of 2 attempts will performed on each subject regardless audible cavitation.
  Arms: Mobilisation; Mobilization with movement
Procedure: Mobilization — The mobilization is a passive oscillatory technique, applied over cervical region in the hypomobile cervical level, the patient will be in prone and the therapist standing at the head of the patients with his thumbs in opposition placed at the level of the facet of the hypomobile cervical vertebra. A posteroanterior(PA) oscillatory pressure is applied, through the thumbs, over the process of the hypomobile vertebra. This oscillatory mobilization, is performed at a frequency of 2Hz (with metronome control/steps) for 2 minutes and repeated 3 times. The rest time between each mobilization was 1 minute.
  Arms: Manipulation group; Mobilization with movement
Procedure: Mobilization with movement — This is a manual therapy technique that consist of applied a sustain pressure over cervical hypomobile symptomatic level and request to patient a pain free movement.
  For performs it, the therapist placed his thumbs on the articular process of that level. The patient sitting. Then, the subject had to perform actively the painful motion while the therapist guides the movement of that vertebra and resists it while returning to neutral. The strength applied was parallel to the plane of the joint, and the procedure was performed in 3 sets of 10 repetitions.
  Arms: Manipulation group; Mobilisation

SUMMARY:
The purpose of this study was to investigate the comparative effectiveness of high velocity and low amplitude (HVLA)vs Mobilization (Mob) vs Mobilization with movement technique (MWMT) in sample of patients with chronic neck pain (CNP). Secondly to evaluate the immediate effects in range of motion and pain thresholds, and the interaction between psychological factors and the outcomes of these three types of manual therapy.

The hypothesis is that all manual therapies techniques will produce similar effects.

DETAILED DESCRIPTION:
The randomized controlled trial included patients with mechanically reproducible CNP, ≥ age 18-years who are randomized into three groups of treatment. The main outcome measures were the Visual Analogue scale (VAS), and, with secondary measures of Neck Disability Index (NDI), Global Rating Of Change (GROC), Cervical Range Of Motion (CROM), Pressure Pain Threshold (PPT), State Trait Anxiety Inventory (STAI-T), Beck depression Inventory (BDI-II), Tampa Scale for Kinesiophobia, Pain Catastrophizing Scale (PCS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Chronic neck pain

Exclusion Criteria:

* Neck pain is associated with whiplash injuries.
* Resting blood pressure greater than 140/90 mmHg.
* Cervical radiculopathy.
* Cervical disc herniation.
* Fibromyalgia syndrome.
* Previous neck surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | The Patients will be followed for 12 weeks after treatment
  visual analogue scale (VAS). Despite being a subjective evaluation, it has been documented in previous studies its reliability and validity and its sensitivity to the clinical changes. For this reason, this scale has been used in numerous clinical trials on neck pains to evaluate the results. The patient places a vertical mark on a flat horizontal line of 10 cm. One extreme is 0 (no pain) and the other extreme is 10 (maximum pain) and it must be a difference of 2 points in the evaluation range to produce minimal improvement which is clinically significant.

SECONDARY OUTCOMES:
Neck disability | The Patients will be followed for 12 weeks after treatment
  The Neck Disability Index (NDI) is an assessment tool used to record the perceived disability in patients with neck pain .It was developed by Howard Vernon from the well-known and validated Oswestry scale for low back pain. The NDI is a self-administered questionnaire with 10 sections. 7 related to activities of daily living, 2 related to pain and 1 with concentration. Each of the sections is scored from 0 to 5, and the total score is expressed as a percentage relative to the maximum possible. The Spanish version was used in this study. This scale offer a high levels of validity and reliability (infraclass correlation coefficient, ICC: 0.88), is stable against different cultural levels and is consistent and reliable. The minimum detectable change is 5 points out of 50, while it is recommended t 7 points as the minimum difference clinically important.
Active Cervical Range of Motion | The Patients will be followed for 12 weeks after treatment
  The ACROM is an instrument that assesses the active range of motion of the cervical segment and has been used in numerous studies to evaluate the results in manual therapy. Furthermore, it has proven to be a reliable method of measuring, providing a range of intra-meter reliability from 0.7 to 0.9 and a range of inter-meter reliability from 0.8 to 0.87. It consists of an inclinometers system. Gravitational inclinometers for flexion-extension and lateral flexion, and magnetic inclinometers for rotation. The patient, sitting in a chair with the goniometer placed over his head, is asked to perform analytical neck movements (flexion, extension, right lateral flexion, left lateral flexion, right rotation and left rotation) to the point of beginning of pain symptoms or, otherwise, to the fullest extent of mobility. Each movement is recorded three times to take the average.
Pressure Pain thresholds (PPTs) | pre-treatment and post-treatment
  Pressure pain threshold (PPT) was used in this study for measure the mechanical hyperalgesia. A digital algometer (FDX 25, Wagner Instruments, Greenwich, CT, USA) comprised of a rubber head (1 cm2) attached to a pressure gauge, was used to measure PPTs. Force was measured in kilograms/f (kgf). The measures were taken 3 times at the cervical spine (C2 spinous process), with an interval of 30 seconds between each of the measurements. An average of the 3 measurements was calculated to obtain a single value for each of the measured points in each of the assessments. The assessor localized the spinous process of C2.

OTHER OUTCOMES:
Satisfaction | The Patients will be followed for 12 weeks after treatment
  The Global Rating Of Change Scale - GROC is also a commonly used scale in clinical research, particularly in patients with neck pain. It is designed to quantify the improvements or deterioration over time, and allows the patient to choose the aspects of life that he considers important. There is variability in the design of the scales, a systematic review in Cochrane quoted seven different designs in the eight studies using a scale of GROC. This scale goes from -7 (much worse) to +7 (much better) with 0 being the midpoint (equally).
Anxiety | pre-treatment
  All participants completed Spanish version 47 of trait subscale of State Trait Anxiety Inventory (STAI-T. The STAI-T has been found to possess adequate reliability (alpha coefficients of 0.93, test-retest reliability of 0.80) and validity.
Depression | pre-treatment
  The level of depressive symptomatology was measured by the Spanish version50 of Beck depression Inventory (BDI-II), a self-report measure which assess affective, cognitive, and somatic symptoms of depression. The BDI has shown good internal consistency both in original sample (alpha coefficient 0.90) and in Spanish population (alpha coefficient 0.92). In addition, both versions has an adequate validity
Kinesiophobia | Pre-treatment
  The Tampa Scale for Kinesiophobia, developed by Miller was used to assess fear of movement and injury. We used the original 17-items version, which has showed good psychometric guarantees.
Catastrophizing | Pre-Treatment
  To evaluate the subject's propensity to catastrophize about pain we used the Spanish version of Pain Catastrophizing Scale (PCS). This scale is a 13-item questionnaire designed to measure the three components of catastrophizing: rumination, magnification and helplessness, resulting this evaluation in a unique score

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez-Carnero, PhD, Principal Investigator — Universidad Europea de Madrid/Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

REFERENCES:
- See also: web site of the University — http://www.urjc.es